CLINICAL TRIAL: NCT00304447
Title: A Phase IV Study of Corticosteroids As Prophylaxis for Infusion-Related Adverse Events to Mylotarg® in Patients With Acute Myelogenous Leukemia (AML)
Brief Title: Study Evaluating the Effect of Corticosteroids on Mylotarg® Infusion-Related Adverse Events in Patients With Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0903X-100863
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Leukemia, Myelocytic, Acute; Infusions, Intravenous
Keywords: Leukemia; Mylotarg; Safety; Adverse Events
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Gemtuzumab

INTERVENTIONS:
Drug: Mylotarg

SUMMARY:
The purpose of this study is to evaluate the effect of corticosteroids on the frequency and severity of Mylotarg® infusion-related adverse events, to evaluate the effect of corticosteroids on the efficacy of Mylotarg® induced complete response (CR) and complete response with incomplete platelet recovery (CRp) at one-month post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD33 positive, resistant or relapsed AML.
* Patients > 18 years of age.
* ECOG performance status 0-2.

Exclusion Criteria:

* Fever (>38), chills or hypotension (systolic BP<105mmHg) in the 48 hours preceding therapy.
* Use of corticosteroids, diphenhydramine or acetaminophen within 24 hours of enrollment.
* Participation in any other Mylotarg® protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-04; Study Completion 2004-01

PRIMARY OUTCOMES:
The effect of corticosteroids on the frequency and severity of Mylotarg® infusion-related adverse events.

SECONDARY OUTCOMES:
The effect of corticosteroids on the efficacy of Mylotarg® induced complete response (CR) and complete response with incomplete platelets recovery (CRp) at one-month post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer